CLINICAL TRIAL: NCT04579939
Title: Oral Glucose Tolerance Testing Using Candy: A Sweet Solution to Improve Screening Compliance in Cystic Fibrosis
Brief Title: Oral Glucose Tolerance Testing Using Candy for Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ana L. Creo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-002446
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): All 10 participants will go through the experimental arm receiving the dextrose candy oral glucose tolerance test.
  Interventions: Diagnostic Test: Candy Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Candy Glucose Tolerance Test — Participants will use a popular dextrose candy alternative to help assess glycemic response.

SUMMARY:
The study aims to determine if a popular dextrose candy alternative yields a similar glycemic curve compared to the standard oral Dextrose solution used in the Oral Glucose Tolerance Test.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 10-21 years.
* Cystic Fibrosis (CF) must be diagnosed.
* Ability to sign informed consent if they are 18 years or older.
* Written parental permission if age 10-17 years old.

Exclusion criteria:

* Active CF flare as determined by the primary CF team .
* Use of steroids.
* Inability to tolerate oral feedings.
* Prior intestinal surgery.
* Concern for allergy or intolerance to dextrose, fructose, or corn derivatives.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Glycemic Response | Baseline, Day 1
  The investigators will obtain glucose values at standard clinical times for oral glucose tolerance testing

SECONDARY OUTCOMES:
Patient and Parent Satisfaction | Day 2
  Self-rated satisfaction using the candy alternative will be assessed via survey

CONTACTS AND LOCATIONS:
Overall Officials: Ana Creo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials